CLINICAL TRIAL: NCT07009847
Title: A Case Control Study to Assess Effectiveness and Safety of The R21/Matrix-M Malaria Vaccine
Brief Title: An Observational Study to Assess Effectiveness and Safety of The R21/Matrix-M Malaria Vaccine
Status: Recruiting | Type: Observational
Sponsor: Serum Institute of India Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: R21-PMS-01
Record Dates: First submitted 2025-04-07; First posted 2025-06-08 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Malaria,Falciparum; Morality
Keywords: clinical malaria; severe malaria; death (all cause)
MeSH Terms: conditions — Malaria, Falciparum; Malaria; Death

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Case control study of Clinical malaria: Clinical Malaria case definition: Presence of axillary temperature ≥ 37.5°C and/ or history of fever within the last 48 hours before the diagnosis is made AND P. falciparum asexual parasitaemia >5000 parasites/μL detected by microscopy.
  This is a case-control study to assess the effectiveness of the R21/Matrix-M Vaccine against clinical malaria in children aged ≥ 5 months of age.
  Surveillance and detection of cases: Cases qualifying the case definitions of clinical, cases will be recruited from the hospitals, clinics or the sub-sites as per the respective case definitions. The required laboratory investigations will be conducted if not already done to ensure the child meets the respective case definition example: e.g. microscopy with parasite density will be conducted in the suspected cases of clinical malaria.
  For clinical malaria cases in high-transmission perennial areas, the ratio of case: control will be 1:1. Controls will be matched for age and neighborhood.
  Interventions: Other: Case control study of clinical malaria
- Case control study of Severe malaria: Severe Malaria case definition: Presence of P. falciparum parasitaemia detected by microscopy AND one or more of the disease severity criteria.
  This is a case-control study to assess the effectiveness of the R21/Matrix-M Vaccine against severe malaria in children aged ≥ 5 months of age. Surveillance and detection of cases: Cases qualifying the case definitions of severe malaria, cases will be recruited from the hospitals, clinics or the sub-sites as per the respective case definitions. The required laboratory investigations will be conducted if not already done to ensure the child meets the respective case definition. For severe malaria cases, the ratio of case: control will be 1:4. Controls will be matched for age and neighborhood.
  Interventions: Other: Case control study of severe malaria
- Case control study of death (all cause): Death (all-cause) case definition: Children who died, of any cause excluding trauma or elective surgery, who were eligible to have received the R21/Matrix-M vaccine based on their date of birth.
  This is a case-control study to assess if the R21 vaccine recipients are at an increased risk due to (all cause) mortality in children aged ≥ 5 months of age. Surveillance and detection of cases: For deaths, cases will be recruited from the hospital or the community (house visits). Cause of death can be ascertained from hospital or available medical records as well as discussions with family or healthcare professionals who may have been involved. For death (all cause) cases, the ratio of case: control will be 1:4. living controls will be enrolled and matched for age and neighborhood.
  Interventions: Other: Case control study of death (all cause)

INTERVENTIONS:
Other: Case control study of clinical malaria — Case control study of clinical malaria
  Groups: Case control study of Clinical malaria
Other: Case control study of severe malaria — Case control study of severe malaria
  Groups: Case control study of Severe malaria
Other: Case control study of death (all cause) — Case control study of death (all cause)
  Groups: Case control study of death (all cause)

SUMMARY:
This is an observational case-control study to assess the effectiveness of the R21/Matrix-M vaccine against severe malaria, clinical malaria (in high transmission perennial areas), and to assess if the R21 vaccine recipients are at an increased risk of deaths (all-cause). Clinical malaria, severe malaria and death (all-cause) cases will be enrolled in study. For each case (severe or death) 4 controls matched for age and neighborhood will be enrolled whereas for clinical malaria case, 1 matched control will be enrolled.

1. Proportion of vaccinated and unvaccinated children amongst Severe Malaria Cases caused by P. falciparum.
2. Proportion of vaccinated and unvaccinated children amongst Clinical Malaria Cases in high-transmission perennial areas caused by P. falciparum.
3. Proportion of vaccinated and unvaccinated children in cases of death (all cause)
4. Exploratory effectiveness endpoint: Proportion of vaccinated and unvaccinated children in the hospitalized clinical and severe malaria cases.

DETAILED DESCRIPTION:
The study will be conducted at multiple centers with the appropriate research infrastructure to carry out safety and/or effectiveness research across different countries where the R21/Matrix-M vaccine is (or will be) approved and deployed for vaccination with subsequent population uptake.

The cases will be enrolled from hospitals/clinics and the matched controls will be recruited from the community by visiting the neighborhood.

Children eligible for receiving R21/Matrix-M vaccine, residing in the geographical area where the vaccine has been deployed will be considered as either cases or controls if they meet the eligibility criteria. All participants will be screened for eligibility after obtaining informed written consent from parents/legal guardians/ caregivers.

Surveillance and detection of cases: Cases qualifying the case definitions of clinical or severe malaria, cases will be recruited from the hospitals, clinics or the sub-sites.

For deaths, cases will be recruited from the hospital or the community. Cause of death will be ascertained from hospital or available medical records as well as discussions with family or healthcare professionals who may have been involved.

Identification of controls: Four controls for each case will be recruited by study physician or field staff from community for severe malaria and death cases. For clinical malaria cases in high-transmission perennial areas, case: control ratio will be 1:1. Controls will be matched for age and neighborhood. Controls should be residing in the same neighborhood as the respective case, but not from the same house. Living controls will be enrolled against the death cases. Vaccination status will be confirmed from the vaccination/immunization cards, hospital/clinic records, home based registers, or national immunization database. History from the parents/ guardians/ caregivers will be considered in case of non-vaccination. Field staff may visit the homes of controls and (if required) cases for collection of the required data.

ELIGIBILITY:
Inclusion Criteria:

For Cases- A male or female child eligible to have received R21/Matrix-M Vaccine based on age. 2 Parent/legal guardian/ caregiver of the child willing to provide the written informed consent for their child's participation in the study.

3 Parent/legal guardian/ caregiver willing to comply with the study requirements and share or allow access to the data regarding the vaccination status and medical records with the study personnel.

4 Resident of the R21/Matrix-M vaccine implementation area and brought to the study hospital /clinic or sub-site with clinical complaints. 5 Child meeting the respective case definition (Severe Malaria, Clinical Malaria or Death due to any cause).

For Controls- A male or female child eligible to have received R21/Matrix-M Vaccine based on age. The matched control should have a date of birth within 60 days of that of the case.

2. Parent/legal guardian/ caregiver of the child willing to provide the informed consent for their child's participation in the study.

3. Parent/ legal guardian/ caregiver willing to comply with the study requirements and share or allow access to the data regarding the vaccination status and medical records with the study personnel 4. Resident of the R21/Matrix-M vaccine implementation area and who would have sought treatment at the same hospital if they had developed symptoms. Resident will be defined as child and/or child's parents/ guardian/caregiver eating and sleeping in a household in the location for most days of the week from past 6 months. The matched control should be residing in the same neighborhood as the respective case, but not from the same household.

Exclusion Criteria:

For Cases-

1. Parent/legal guardian/ caregiver not consenting to let the child participate or not permitting to access the data related to vaccination or other medical records.
2. Child not meeting the respective case definition (Severe Malaria, Clinical Malaria or Death due to any cause).
3. Received one or more doses of RTS,S/AS01 vaccine in the past.

For Controls-

1. Parent/legal guardian/ caregiver not consenting to let the child participate or not permitting to access the data related to vaccination or other medical records.
2. Child meeting any of the case definitions (Severe Malaria, Clinical Malaria).
3. Child having history suggestive of clinical malaria in past 30 days (applicable for clinical malaria and severe malaria case-control studies only).
4. Received one or more doses of RTS,S/AS01 vaccine/s in the past.

Min Age: 5 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population will comprise children aged 5 months and above who live in R21-Malaria vaccine implementation areas in Uganda, Burkina Faso, Nigeria, Cote d'ivoire and who were eligible to have received R21-malaria vaccine based on their date of birth and age
Sampling Method: Non-Probability Sample
Enrollment: 2308 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Vaccine Effectiveness against Severe Malaria caused by P. falciparum | through study, an average of one year
  Proportion of vaccinated and unvaccinated children amongst Severe Malaria Cases caused by P. falciparum.
Vaccine Effectiveness against clinical malaria caused by P. falciparum in high perennial transmission areas | through study, an average of one year
  Proportion of vaccinated and unvaccinated children amongst Clinical Malaria Cases caused by P. falciparum.
Risk of death (all cause) due to R21-vaccination | through study, an average of one year
  Proportion of vaccinated and unvaccinated children in cases of death

CONTACTS AND LOCATIONS:
Locations (5):
- Unité de Recherche Clinique de Nanoro (URCN), Institut de Recherche en Sciences de la Santé, Direction Régionale du Centre-Ouest (IRSS-DRCO), Bousse, Boussé, Burkina Faso, Burkina Faso
- Centre de Recherche et de Lutte contre le Paludisme Institut National de Santé Publique, boulevard Nangui Abrogoua près État Major des Armées, Toumodi, Côte d’Ivoire
- University of Ilorin Department of Pediatrics University of Ilorin Teaching Hospital, Ilorin, Nigeria, Yenagoa, Bayesla, Nigeria
- Uganda (2):
  - Infectious Diseases Research Collaboration (IDRC), Uganda, Busia, Uganda
  - Makerere University College of Health Sciences, Mukono

IPD SHARING:
Plan to Share IPD: Undecided